CLINICAL TRIAL: NCT01608178
Title: Succinic Semialdehyde Dehydrogenase Deficiency: Physiological Markers of Taurine Therapy
Brief Title: Taurine Therapy for SSADH Deficiency
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120123; 12-N-0123
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-12-16

CONDITIONS: Succinic Semialdehyde Dehydrogenase
Keywords: Pediatric Neurotransmitter Disorders; Succinic Semialdehyde Dehydrogenase; GABA; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Succinic semialdehyde dehydrogenase (SSADH) deficiency is a rare genetic disease that results in changes to certain brain chemicals. These chemicals may affect brain excitability, or how likely nerve cells are to turn on. Changes in brain excitability may help to explain the symptoms of the disease, including learning and memory problems, seizures, and poor balance. A supplement called taurine may help people with SSADH deficiency by working on the brain chemical GABA. GABA helps to regulate brain activity. Researchers want to see if taurine can help people with SSADH deficiency.

Objectives:

- To learn more about how taurine affects the brain in people with SSADH deficiency.

Eligibility:

- Individuals at least 12 years of age who have SSADH deficiency.

Design:

* Participants will be screened with a physical exam and medical history. They will provide blood and urine samples. They will also take taurine supplements as part of this protocol.
* Participants will have two sets of study tests. One set will be given while participants are taking taurine. The second will be given when they are not taking it. Each testing session will take about 2 days to complete.
* Half of the participants will have the "off taurine" testing before starting on the taurine supplement. The other half will start taking taurine first, have the "on taurine" testing, and have the "off taurine" testing about 3 months after stopping taurine. Participants may decide the order in which they will have the testing done.
* Participants will have the following tests at the two test visits:
* Paper and pencil tests of learning and memory.
* Transcranial magnetic stimulation to study the excitability of nerve cells.
* Imaging studies to show GABA receptors in the brain and measure their activity.
* Electroencephalogram to measure brain waves.
* Lumbar puncture to collect spinal fluid.
* Participants will be monitored with regular study visits while they receive the taurine supplement treatment.

DETAILED DESCRIPTION:
Objective: To study the physiologic effects of taurine therapy in patients with succinic semialdehyde Dehydrogenase (SSADH) deficiency.

Study Population: Eighteen children and adults with SSADH deficiency receiving taurine.

Design: This small open label trial will evaluate the effect of taurine treatment on key SSADH biomarkers and neurocognitive performance. Study evaluations will include neurological and neuropsychological examinations, positron emission tomography (PET) with 11C-flumazenil (FMZ), (optional and only for those over age 18), magnetic resonance spectroscopy (MRS) (optional) and cerebrospinal fluid (CSF) collection (optional) to measure gamma-aminobutyric acid (GABA) levels, and transcranial magnetic stimulation (TMS) to measure cortical excitation and inhibition, in patients given taurine for SSADH deficiency.

The evaluations will be performed twice, on and off therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Persistent 4-hydroxybutyric aciduria (gamma-hydroxybutyric aciduria).

Documented succinic semialdehyde dehydrogenase enzyme deficiency.

Patients will be at least 12 years old.

Be enrolled in the taurine study at CNMC.

EXCLUSION CRITERIA:

Pregnancy or lactation.

Patients with a history of other significant medical disorders.

Patients requiring treatment with drugs known to affect the GABAergic system, including vigabatrin, barbiturates, and benzodiazepines.

Hearing loss. The effect of TMS on hearing is not fully known. Patients will be screened with an Audiometer.

Abnormal platelets or coagulation studies suggesting increased risk for lumbar puncture or TMS

Exclusions for MRI and MRS: pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, or shrapnel fragments, welders and metal workers.

Exclusions for TMS: people with implanted medical devices such as pacemakers, implanted pumps, stimulators, or cochlear implants or in people who have metal objects inside the eye or skull.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-04-27; Study Completion 2013-12-16

PRIMARY OUTCOMES:
TMS parameters of cortical excitation and inhibition.

SECONDARY OUTCOMES:
Change in CSF GABA, GHB, succinic semialdehyde, homocarnosine, 4,5-dihydroxyhexanoic acid, D-2-hydroxyglutaric acid, homovanillic acid, and 5-HIAA levels.

CONTACTS AND LOCATIONS:
Overall Officials: William H Theodore, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Al-Essa MA, Bakheet SM, Patay ZJ, Powe JE, Ozand PT. Clinical, fluorine-18 labeled 2-fluoro-2-deoxyglucose positron emission tomography (FDG PET), MRI of the brain and biochemical observations in a patient with 4-hydroxybutyric aciduria; a progressive neurometabolic disease. Brain Dev. 2000 Mar;22(2):127-31. doi: 10.1016/s0387-7604(99)00121-7. PMID 10722966
- [Background] Arnulf I, Konofal E, Gibson KM, Rabier D, Beauvais P, Derenne JP, Philippe A. Effect of genetically caused excess of brain gamma-hydroxybutyric acid and GABA on sleep. Sleep. 2005 Apr;28(4):418-24. doi: 10.1093/sleep/28.4.418. PMID 16171286
- [Background] Simmons FB. Letter: Stellate ganglion blocks for idiopathic sensorineural hearing loss. Arch Otolaryngol. 1976 Jun;102(6):384-5. doi: 10.1001/archotol.1976.00780110096021. No abstract available. PMID 1275811